CLINICAL TRIAL: NCT02755181
Title: Assessment of Longitudinal Functional Magnetic Resonance Imaging (fMRI) as a Brain Measure for Impulsivity in a Borderline Personality Disorder (BPD) Model
Brief Title: fMRI in Impulsivity
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 352.2067
Record Dates: First submitted 2016-04-08; First posted 2016-04-28 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Impulse Control Disorders; Borderline Personality Disorder
MeSH Terms: conditions — Disruptive, Impulse Control, and Conduct Disorders; Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- BPD: Borderline Personality Disorder as diagnosed by DSM-5
  Interventions: Behavioral: Experimental
- normal volunteers: normal volunteers
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Experimental — with functional imaging and behavioural measurements at baseline and 4 weeks

SUMMARY:
This study aims to use resting-state and task based functional Magnetic Resonance Imaging (fMRI) as a tool to evaluate trait characteristics of impulsivity in subjects with borderline personality disorder.

ELIGIBILITY:
Inclusion criteria:

* Healthy Controls: Volunteers (age 18-50 yrs) in generally good Psychiatric and non-Psychiatric medical health
* Borderline Personality Disorder subjects: Research volunteers (age 18-50 yrs) who meet DSM-5 criteria for Borderline Personality Disorder

Exclusion criteria:

All Participants:

* Current medications which affect the central nervous system or vascular activity, such as anti-depressants, anxiolytics, or blood-pressure medications
* Positive urine drug screen for cocaine, opioids, amphetamine, and benzodiazepines
* Positive breathalyzer test for alcohol
* History of clinically significant neurologic disorders or head trauma with loss of consciousness greater than 30 minutes
* Clinically significant non-psychiatric medical disorder requiring ongoing treatment.
* Unwillingness or inability to sign a written informed consent form
* Pregnancy as assessed by a urine test for ß-HCG at each visit
* Medical or physical contraindications for participation based on medical history interview, labs, and physical exam
* Metal fragments or other bodily metal (e.g., pacemaker, orthopedic prosthesis),claustrophobia, or any other condition that would put the subjects at risk for MRI scanning

In addition, Healthy Controls excluded, if:

* DSM-5 diagnoses of Personality Disorders (based on SCID-II)
* DSM-5 diagnoses based on the SCID-I (including the eating disorders module)
* History of arrest or incarceration

In addition, Borderline Personality Disorder Subjects excluded if:

* DSM-5 diagnoses
* DSM-5 Personality Disorder other than Cluster B Personality disorders
* Current psychoactive medications
* Further exclusion criteria apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: BPD and normal volunteers
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2016-07-22 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Affective Faces Task (AFT) fMRI response | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Monetary Incentive Delay (MID) fMRI task response | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for resting-state functional magnetic resonance imaging (fMRI) activity | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Go/ No Go functional magnetic resonance imaging (fMRI) response | up to 5 weeks

SECONDARY OUTCOMES:
Change from baseline to 4 week follow-up visit for Eye Tracking | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Immediate Memory Task (IMT) behavioral test | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Computerized monetary choice procedure behavioral test | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Stop-signal paradigm behavioral test | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Barratt Impulsiveness Scale v.11 (BIS-11) | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Profile of Mood States behavioral test | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Go/ No Go task behavioral test | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Urgency, Premeditation, Perseverance, Sensation Seeking, and Positive Urgency (UPPS-P) Impulsive behavior Scale, subscale for premeditation | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Urgency, Premeditation, Perseverance, Sensation Seeking, and Positive Urgency (UPPS-P) Impulsive behavior Scale, subscale for perseverance | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Urgency, Premeditation, Perseverance, Sensation Seeking, and Positive Urgency (UPPS-P) Impulsive behavior Scale, subscale for sensation seeking | up to 5 weeks
Stability in scores measured as change from baseline to follow-up visit at 4 (+/-1) weeks for Urgency, Premeditation, Perseverance, Sensation Seeking, and Positive Urgency (UPPS-P) Impulsive behavior Scale, subscale for urgency | up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States